CLINICAL TRIAL: NCT00714467
Title: Expert System and Family Assisted Interventions for Chinese Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TURSG-03-102-01 PBP; ACS Grant: TURSG-03-102-01 PBP; H10315-21203-07
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; Asian; Chinese American; family support; social support; stage-based intervention
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Expert system (stage-based manual and 3 individualized tailored feedback reports) only for smokers, paired-supporters (family or friend participant) do not receive any study intervention
  Interventions: Behavioral: Expert System Only
- 2 (Experimental): Expert system (stage-based manual and 3 individualized tailored feedback report) to all the smoker participants; a family assisted intervention in a form of a self-help booklet that discusses specific strategies to work with smokers at each stage of change to the paired-supporters
  Interventions: Behavioral: Family Assisted

INTERVENTIONS:
Behavioral: Expert System Only — expert system intervention only to the smoker participants which includes a stage-based manual and a series of 3 individualized tailored feedback report at baseline, 3, and 6 months. The paired-supporters receive assessments only and no intervention.
  Arms: 1
Behavioral: Family Assisted — The smoker participants received an expert system intervention (same intervention for those in the Expert system intervention) which includes a stage-based manual and a series of 3 individualized tailored feedback report at baseline, 3, and 6 months. The paired-supporters will receive a a self-help booklet based on the Transtheoretical Model of Change (TTM) that will aim at teaching the supporters how to use the stages of change framework to apply different strategies that best match with smokers' readiness to quit smoking.
  Arms: 2

SUMMARY:
In this study, we choose to specifically recruit Chinese, the largest ethnic group of the Asian and Pacific Islander community,2 as an initial step to increase our understanding of the role of family or supportive others in the process of smoking cessation among Asian Americans. We propose the following specific aims for the study:

1. Examine the effectiveness of proactive recruitment of Chinese smokers into a smoking cessation treatment program through their family or friends.
2. Test the efficacy of a family assisted intervention using the stages of change approach in promoting smoking cessation in the context of an expert system intervention.
3. Explore the role of supportive and non-supportive behaviors in relation to both short-term and long-term smoking cessation outcomes in the presence of the expert system intervention.

DETAILED DESCRIPTION:
Limited empirical data are available on effective intervention approaches targeting Chinese American smokers. The overall goal of this study is to increase our understanding of the role of family or social support in the facilitation of the process of smoking cessation among Chinese smokers. We propose the following specific aims for the study: 1) Examine the effectiveness of proactive recruitment of Chinese smokers into a smoking cessation treatment program through their family or friends; 2) Test the efficacy of a family assisted intervention using the stages of change approach in promoting smoking cessation in the context of an expert system intervention; 3) Explore the role of supportive and non-supportive behaviors in relation to both short-term and long-term smoking cessation outcomes in the presence of the expert system intervention. This study will develop a family-assisted intervention in the form of a self-help booklet based on the Transtheoretical Model of Change (TTM) that will aim at teaching the supporters how to use the stages of change framework to apply different strategies that best match with smokers' readiness to quit smoking. This study will conduct focus groups and a pilot study to pre-test the study intervention and study procedures. The main randomized trial will recruit a total of 800 supporters and 800 smokers who are ethnic Chinese residing in the State of California. Each supporter-smoker pair will be randomly assigned to either 1) the expert system intervention only or 2) the expert system plus family-assisted intervention condition after baseline assessment by mail. All smokers in either condition will receive the expert system intervention. Half of the supporters will receive family-assisted intervention materials. All participants will be assessed at baseline, 3, 6, 12, and 18 months by mail or telephone. It is hypothesized that the expert system plus family-assisted intervention condition will yield significantly higher abstinence rates and higher portions to report quit attempts at follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* self-identified ethnic Chinese
* men and women
* above age 18
* can read and speak Chinese or English
* reside in the State of California at baseline
* to participate as a supporter, the participant must have a targeted smoker who meet the smoker eligibility criteria who provides consent to participate in the study as a smoker participant
* to participate as a smoker, the participant must have smoked at least 100 cigarettes in lifetime and have smoked at least 5 cigarettes in the past 7 days, and have a supporter who provides consent to be a supporter participant

Exclusion Criteria:

* smoker participant currently engage in other smoking cessation programs or efforts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1280 (Actual)
Dates: Start 2004-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
self-report 7-day smoking abstinence | 12 months, 18 months

SECONDARY OUTCOMES:
self-report of at least a 24-hour quit attempt | 12 months, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Janice Tsoh, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Langley Porter, San Francisco, California, United States

REFERENCES:
- [Background] Luk JW, Tsoh JY. Moderation of gender on smoking and depression in Chinese Americans. Addict Behav. 2010 Nov;35(11):1040-3. doi: 10.1016/j.addbeh.2010.06.021. Epub 2010 Jun 25. PMID 20655665